CLINICAL TRIAL: NCT04578782
Title: Pilot Study for the Evaluation of the Efficacy of OnabotulinumtoxinA in High Frequency Migraine
Brief Title: Efficacy of OnabotulinumtoxinA in Migraine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: IRCCS National Neurological Institute "C. Mondino" Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FM-BOEM
Record Dates: First submitted 2020-10-01; First posted 2020-10-08 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-09

CONDITIONS: Migraine
Keywords: Migraine; OnabotulinumtoxinA
MeSH Terms: conditions — Migraine Disorders | interventions — Botulinum Toxins, Type A; incobotulinumtoxinA

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BOTOX (Experimental): 155 UI of Botox were injected according to the approved PREEMPT protocol (the only FDA-approved injection pattern for chronic migraine), in 31 sites. From visit 5, the PREEMPT 'follow-the-pain' paradigm was applied in patients falling in the 'non-responder' or 'partial responder' classes after the first BoNT-A injection, with the possibility to increase the doses up to 195 UI in maximum 39 sites. The injections were every 3 months for 4 cycles
  Interventions: Drug: OnabotulinumtoxinA

INTERVENTIONS:
Drug: OnabotulinumtoxinA — BOTOX contains onabotulinumtoxinA, an acetylcholine release inhibitor and a neuromuscular blocking agent available in the lyophilized form of purified clostridium botulinum toxin type A, suitable for injection, for intramuscular, intradetrusor, or intradermal use. The recommended dilution is 100 Units/2 mL, with a final concentration of 5 Units per 0.1 mL. The recommended dose for treating chronic migraine is 155 Units administered intramuscularly using a sterile 30-gauge, needle as 0.1 mL (5 Units) injections per each site.
  Other Names: BonT-A (Botox®)

SUMMARY:
Population studies estimate that patients who have episodic migraine transition to chronic migraine at a rate of about 2.5% per year.

CM is a devastating disorder associated to severe disability. Patients with CM frequently overuse symptomatic medications in the attempt to control their disease, which adds up to the high costs associated to the disorder In this frame, it seems of the outmost importance to strive at preventing the transition from EM to CM.

At the moment Onabotulinum toxin A (BoNT-A) represents the only drug specifically approved for CM prophylaxis.

The aim of the present study was to evaluate the efficacy of BoNT-A in reducing the number of migraine days in a population of migraineurs with a high frequency of migraine attacks over a 12-month period.

DETAILED DESCRIPTION:
Episodic migraine (EM) is a common type of disabling headache that affects up to 15% of the general population. In a minority of patients, migraine progressively increase in frequency, until it becomes chronic. According to the criteria of the International Headache Society chronic migraine (CM) is characterized by a headache that is present on at least 15 days per month over at least three months period, with migraine characteristics on at least 8 days/month. Population studies estimate that patients who have episodic migraine transition to chronic migraine at a rate of about 2.5% per year.

CM is a devastating disorder associated to severe disability. Patients with CM frequently overuse symptomatic medications in the attempt to control their disease, which adds up to the high costs associated to the disorder In this frame, it seems of the outmost importance to strive at preventing the transition from EM to CM.

Transition to CM rarely is a rapid phenomenon. Most often it occurs over several months or years during which the frequency of attacks progressively increases as does the intake of acute medications. High monthly headache frequency is a risk factor for the progression of episodic migraine to chronic migraine. Compelling evidence from clinical and pre-clinical studies suggests that the transformation into CM is associated to, and probably brought about by, plastic changes in the peripheral and central nervous system induced by the repetitive occurrence of pain attacks. These changes configure a condition of chronic sensitization, usually associated to a reduced response to treatments.

In this frame, it is noteworthy that the investigators previously showed that patients with CM overusing acute medications bear a condition of enhanced facilitation of spinal cord pain processing that is detectable with specific neurophysiological evaluations. The situation normalizes, i.e. pain facilitation is reduced, 60 days after successful treatment. Similarly, the Danish group showed that patients with chronic headache associated to medication overuse (most of whom were suffering from CM) are sensitized to pain, and pain perception continues to normalise over a period of at least 12 months when patients are successfully treated.

At the moment Onabotulinum toxin A (BoNT-A) represents the only drug specifically approved for CM prophylaxis.

Seven different subtypes of botulinum toxin (A-G) are known. A highly-diluted preparation of botulinum toxin type A was introduced in clinical practice in the 1970s and 1980s to treat squint and blepharospasm. Since then, it has found uses in other areas of medicine including dystonia (including writer's cramp), post-stroke spasticity, and hyperhidrosis but in the mid-1990s a number of people reported improvement in headaches in patients receiving botulinum toxin for other reasons. Finally, in the first decade of 2000 two trials, the Phase 3 Research Evaluating Migraine Prophylaxis Therapy (PREEMPT) recruited 1384 patients with chronic migraine, and randomised them to treatment with BoNT-A (Botox® by Allergan Industries) or placebo. These patients were suffering on average 20 days of headache each month, of which 18 were moderate or severe. Those randomised to Botox®® received fixed-site, fixed dose injections every 12 weeks over 56 weeks. These injections covered seven specific areas of the head and neck, with a total dose of between 155-195 units. At six months, after two cycles of treatment, those treated with Botox® had on average eight less days of headache each month. After 12 months, 70% of those treated had ≤50% the number of headaches that they had done originally. Botox® was well-tolerated, the commonest side effects being neck pain (6.7%), muscular weakness (5.5%), and drooping of the eyelid (3.3%). No serious irreversible side effects have ever been reported in trials of Botox® in headache.

These studies led in 2013 to the approval by AIFA of Botox® as a drug form CM prophylaxis.

An increasing body of evidence suggests that BoNT-A acts on peripheral trigeminal endings by inhibiting the release of nociceptive neuropeptides - such as calcitonin gene-related peptide (CGRP) - and glutamate, as well as the expression of the transient receptor potential vanilloid 1, thereby reducing directly peripheral sensitization, and, indirectly, central sensitization. It is noteworthy that preclinical data also suggest a central antinociceptive action for BoNT-A, probably associated with an enhanced opioidergic and GABA-ergic transmission.

Taken together, these observations provide the rationale of this study, which is to evaluate whether BoNT-A treatment is effective in reducing the number of migraine days in migraineurs with a high monthly frequency of migraine attacks.

This study is a phase II, single group, non-randomized, non-controlled, open label trial performed at a single centre: Mondino Foundation.

Patients affected by migraine with high frequency of attacks per month were enrolled at the Headache Science Centre of IRCCS C. Mondino in Pavia. After the screening visit, selected patients were evaluated with a headache daily diary for a period of 1 month. If the diagnosis of episodic migraine with high frequency of attacks per month was confirmed, the patient were enrolled and received the treatment with BoNT-A at the centre every 3 months for 4 cycles (at visit V2-V5-V8-V11). At the first administration of the treatment (V2), 155 UI of Botox were injected according to the approved PREEMPT protocol, in 31 sites. From visit 5, the PREEMPT 'follow-the-pain' paradigm will be applied in patients falling in the 'non-responder' or 'partial responder' classes after the 1st BoNT-A injection, with the possibility to increase the doses up to 195 UI in maximum 39 sites.

Every 3 month the patients were asked to fill in 3 validated questionnaires for the quantification of disability (Migraine Disability Assessment Score Questionnaire - MIDAS), quality of life (Mental Status Questionnaire - MSQ), anxiety and depression (Hospital Anxiety and Depression Scale - HADS). Every month the patient also received a phone call from the site personnel in order to be updated on the clinical conditions.

During all the study period the patient was asked to complete a daily headache diary in order to evaluate the clinical condition and the medications use.

ELIGIBILITY:
Inclusion Criteria:

* Subjects fulfilling the diagnostic criteria for migraine without or with aura of the International Headache Classification with a number of migraine days ranging from 9 to 14 days/month in the previous 3 months.
* The frequency needs to be confirmed over the 28 days before the screening visit .
* Subjects have to be in general good health, as confirmed by medical history, baseline physical examination, baseline neurological exam and vital signs.
* Females have to be postmenopausal for at least one year, surgically sterile or otherwise incapable of pregnancy, or using an acceptable method of birth control.

Exclusion Criteria:

* Previous failure of more than two adequate trials of medications from different drug classes used for migraine prophylaxis;
* Onset of migraine after age 50;
* Exclusively migraine aura without headache;
* Diagnosis of other primary or secondary headache disorders. Episodic tension-tyep headache is allowed if the patient can distinguish clearly between attack of migraine and of tension-type headache;
* Another chronic painful condition (e.g. osteoarthritis, low back pain);
* A significant medical history or medical condition of neurological, cardiovascular hepatic or renal disease;
* History of suicide attempt or suicidal ideation or of a major psychiatric disorder;
* History of drug or alcohol abuse within the past two years.
* Known hypersensitivity to botulinum toxin type A or to any of the other ingredients used to form 'Botox®'

Withdrawal criteria

• Severe side effects, diary completion insufficient for evaluation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2018-03-13 (Actual); Primary Completion 2020-05-31 (Actual); Study Completion 2020-05-31 (Actual)

PRIMARY OUTCOMES:
Migraine days/month | In the last 16 weeks of the study period as compared to the 4 baseline weeks.
  To evaluate the efficacy of BoNT-A in reducing the number of migraine days in a population of migraineurs with a high frequency of migraine attacks over a 12-month period.
  Based on the response in terms of percent reduction of migraine days from baseline, the following classes will be identified:
  * non-responders: reduction < 30%;
  * partial responders: reduction ranging from 30 to 49%;
  * responders: reduction ranging from 50% to 74%;
  * optimal responders: reduction >75%.

SECONDARY OUTCOMES:
Monthly headache days | In the last 16 weeks of the study period as compared to the 4 baseline weeks.
  To evaluate the efficacy of BoNT-A in a population of migraineurs with a high frequency of migraine attacks over a 12-month period.
Migraine attack intensity | In the last 16 weeks of the study period as compared to the 4 baseline weeks.
  To evaluate the efficacy of BoNT-A in a population of migraineurs with a high frequency of migraine attacks over a 12-month period.
Monthly use of acute drugs | In the last 16 weeks of the study period as compared to the 4 baseline weeks.
  To evaluate the efficacy of BoNT-A in a population of migraineurs with a high frequency of migraine attacks over a 12-month period.
Migraine Disability Assessment Score Questionnaire (MIDAS) | In the last 16 weeks of the study period as compared to the 4 baseline weeks.
  To evaluate disability in a population of migraineurs with a high frequency of migraine attacks over a 12-month period.
  The MIDAS questionnaire is a 7-item questionnaire (with 5 scored items) designed to measure headache-related disability, to improve physician-patient communication, and to identify patients with high treatment needs. Higher values are worse outcomes.
Mental Status Questionnaire (MSQ) | In the last 16 weeks of the study period as compared to the 4 baseline weeks.
  To evaluate the quality of life in a population of migraineurs with a high frequency of migraine attacks over a 12-month period.
  The MSQ is a 10-item questionnaire, which provides a brief, objective, and quantitative measurement of cognitive functioning of elderly people.
Hospital Anxiety and Depression Scale (HADS) | In the last 16 weeks of the study period as compared to the 4 baseline weeks.
  To evaluate levels of anxiety and depression in a population of migraineurs with a high frequency of migraine attacks over a 12-month period.
  The HADS is commonly used by doctors to determine the levels of anxiety and depression that a person is experiencing. The HADS is a fourteen item scale that generates: Seven of the items relate to anxiety and seven relate to depression. Each item on the questionnaire is scored from 0-3, with three denoting highest anxiety or depression level.

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Tassorelli, MD, Principal Investigator — Headache Science Center
Locations (1):
- Headache Science Center, Pavia, Italy

REFERENCES:
- [Background] Bigal ME, Serrano D, Buse D, Scher A, Stewart WF, Lipton RB. Acute migraine medications and evolution from episodic to chronic migraine: a longitudinal population-based study. Headache. 2008 Sep;48(8):1157-68. doi: 10.1111/j.1526-4610.2008.01217.x. PMID 18808500
- [Background] Katsarava Z, Schneeweiss S, Kurth T, Kroener U, Fritsche G, Eikermann A, Diener HC, Limmroth V. Incidence and predictors for chronicity of headache in patients with episodic migraine. Neurology. 2004 Mar 9;62(5):788-90. doi: 10.1212/01.wnl.0000113747.18760.d2. PMID 15007133
- [Background] Bigal ME, Rapoport AM, Sheftell FD, Tepper SJ, Lipton RB. Chronic migraine is an earlier stage of transformed migraine in adults. Neurology. 2005 Nov 22;65(10):1556-61. doi: 10.1212/01.wnl.0000184477.11569.17. PMID 16301481
- [Background] Lai TH, Protsenko E, Cheng YC, Loggia ML, Coppola G, Chen WT. Neural Plasticity in Common Forms of Chronic Headaches. Neural Plast. 2015;2015:205985. doi: 10.1155/2015/205985. Epub 2015 Aug 20. PMID 26366304
- [Background] Perrotta A, Arce-Leal N, Tassorelli C, Gasperi V, Sances G, Blandini F, Serrao M, Bolla M, Pierelli F, Nappi G, Maccarrone M, Sandrini G. Acute reduction of anandamide-hydrolase (FAAH) activity is coupled with a reduction of nociceptive pathways facilitation in medication-overuse headache subjects after withdrawal treatment. Headache. 2012 Oct;52(9):1350-61. doi: 10.1111/j.1526-4610.2012.02170.x. Epub 2012 Jun 1. PMID 22670561
- [Background] Munksgaard SB, Bendtsen L, Jensen RH. Modulation of central sensitisation by detoxification in MOH: results of a 12-month detoxification study. Cephalalgia. 2013 May;33(7):444-53. doi: 10.1177/0333102412475235. Epub 2013 Feb 21. PMID 23431023
- [Background] Aurora SK, Dodick DW, Turkel CC, DeGryse RE, Silberstein SD, Lipton RB, Diener HC, Brin MF; PREEMPT 1 Chronic Migraine Study Group. OnabotulinumtoxinA for treatment of chronic migraine: results from the double-blind, randomized, placebo-controlled phase of the PREEMPT 1 trial. Cephalalgia. 2010 Jul;30(7):793-803. doi: 10.1177/0333102410364676. Epub 2010 Mar 17. PMID 20647170
- [Background] Diener HC, Dodick DW, Aurora SK, Turkel CC, DeGryse RE, Lipton RB, Silberstein SD, Brin MF; PREEMPT 2 Chronic Migraine Study Group. OnabotulinumtoxinA for treatment of chronic migraine: results from the double-blind, randomized, placebo-controlled phase of the PREEMPT 2 trial. Cephalalgia. 2010 Jul;30(7):804-14. doi: 10.1177/0333102410364677. Epub 2010 Mar 17. PMID 20647171
- [Derived] Martinelli D, Arceri S, De Icco R, Allena M, Guaschino E, Ghiotto N, Bitetto V, Castellazzi G, Cosentino G, Sances G, Tassorelli C. BoNT-A efficacy in high frequency migraine: an open label, single arm, exploratory study applying the PREEMPT paradigm. Cephalalgia. 2022 Feb;42(2):170-175. doi: 10.1177/03331024211034508. Epub 2021 Aug 18. PMID 34404257